CLINICAL TRIAL: NCT04346836
Title: Low-intensity Exercise as a Predictor of Mental Health in Women With Metabolic Syndrome
Brief Title: Low-intensity Exercise in Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wroclaw University of Health and Sport Sciences (Other)
Collaborators: Foundation for Senior Citizen Activation SIWY DYM (Other)
Responsible Party: Principal Investigator, Joanna Szczepańska-Gieracha, Professor, Wroclaw University of Health and Sport Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 59/0203/S/04
Record Dates: First submitted 2020-04-09; First posted 2020-04-15 (Actual); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: Metabolic Syndrome; Obesity; Hypertension; Hyperlipidemias; Glucose Metabolism Disorders
Keywords: metabolic syndrome; low-intensity exercise; mental health; depression; stress; physical activity; women
MeSH Terms: conditions — Metabolic Syndrome; Obesity; Hypertension; Hyperlipidemias; Glucose Metabolism Disorders; Psychological Well-Being; Depression; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metabolic Syndrome (Experimental): Elderly women with Metabolic Syndrome
  24 sessions of low-intensity exercise and psychoeducation, twice a week over 12 weeks.
  Interventions: Behavioral: Low-intensity, general-fitness exercises; Behavioral: Psychoeducation
- Non-Metabolic Syndrome (Experimental): Elderly women without Metabolic Syndrome.
  24 sessions of low-intensity exercise and psychoeducation, twice a week over 12 weeks.
  Interventions: Behavioral: Low-intensity, general-fitness exercises; Behavioral: Psychoeducation

INTERVENTIONS:
Behavioral: Low-intensity, general-fitness exercises — 24 session of low-intensity, general-fitness exercises (12 weeks, twice a week)
  A single session of exercise lasted 40 minutes and consisted of 42 low-intensity, general-fitness exercises. Perception of effort was monitored using the Borg 6-20 rating the perceived exertion (RPE).
  Thirty-three exercises were done sitting down, seven standing, and two in the hand-and-knees position. The exercises were classified as either aerobic, musculo-articular, or stabilising. The aerobic portion served as a general warm-up for the subsequent exercises, and the musculo-articular section focused on strengthening muscles and enhancing the mobility of joints in the upper limbs, the lower limbs and the torso. Stabilising exercises were designed to improve the stability of the body and to augment spatio-visual coordination.
Behavioral: Psychoeducation — A psychoeducation provided by psychotherapist. Twenty minutes of psychoeducation, which contained mini lectures about mental well-being, psychohygiene and healthy dietary habits.

SUMMARY:
People with metabolic syndrome (MetS) are characterized by a lower quality of life in terms of reduced vital activity, emotional state, and social functioning. Therefore, the investigator's aim was to determine the impact of low-intensity exercise and psychoeducation on depression symptoms and self-perceived stress in women with MetS.

DETAILED DESCRIPTION:
Metabolic syndrome (MetS) is currently one of the major threats to health in highly developed societies. A recent study has demonstrated that depression may be significantly associated with MetS in people aged 60 years or over. The more components of MetS that are evident in the individual, the more depressive symptoms this individual is likely to exhibit.

MetS treatment is essentially founded on implementing lifestyle changes which involve regular physical activity and healthy dietary habits. Systematically undertaking exercise has a beneficial influence on health, particularly on cardiovascular system functions as well as the quality of life and depression status in middle-aged and older women with MetS.

Previous work has shown moderate or high intensity exercise to be optimal for the treatment of MetS. Nevertheless, many patients with MetS have hypertension and obesity. Therefore, for safety reasons, the patient's condition during intensive group exercises should be constantly monitored by a physician or specialized equipment, which generates costs and may limit the availability of this type of intervention.

Hence, the investigator's aim was to determine the impact of 12 weeks of low-intensity exercise, combined with psychoeducation, on the severity of depression symptoms and self-perceived stress in women with MetS.

ELIGIBILITY:
Inclusion Criteria:

The presence of Metabolic Syndrome diagnosed using the International Diabetes Federation-recommended criteria (2006):

* "mandatory" central obesity (defined as waist circumference ≥ 80 cm in females),

and any two of the following:

* raised triglycerides (>150 mg/dL),
* reduced HDL cholesterol (50 mg/dL in females),
* elevated blood pressure (BP; systolic BP > 130 or diastolic BP > 85 mm Hg) ,
* increased fasting plasma glucose (>100 mg/dL),

Exclusion Criteria:

* disturbed cognitive functions (Mini-Mental State Examination > 23),
* the inability to move independently or a motor disability precluding exercise,
* serious neurological or orthopaedic conditions (e.g., advanced Parkinson's disease, severe stroke consequences),
* attending fewer than 13 intervention sessions.

Ages: 60 Years to 85 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2018-05-06 (Actual); Primary Completion 2019-05-10 (Actual); Study Completion 2020-01-10 (Actual)

PRIMARY OUTCOMES:
Change in depression level from baseline | At baseline and after 24 sessions of low-intensity exercise and psychoeducation (week 12)
  As a primary outcome measure, the Geriatric Depression Scale (GDS) was used. GDS is a self-report 15-items measure of well-being and mood in older adults. The patient responds in a "Yes/No" format. Scoring ranges from 0 to 15. A score greater than 5 points is suggestive of depression, and 10 points or more is almost always indicative of depression. With the sensitivity standing at 92%, the GDS is useful in the diagnosis of late-life depression in primary care

SECONDARY OUTCOMES:
Change in perception of stress from baseline | At baseline and after 24 sessions of low-intensity exercise and psychoeducation (week 12)
  As a secondary outcome measure, the Perception of Stress Questionnaire (PSQ) was used. PSQ is a 27-item scale scoring from 1 to 5 for each item. 21 items examine the level of stress in the area of emotional tension, external stress and intrapsychic stress, and 6 items refer to the lie scale. The global scoring for perception of stress ranges from 21 to 105 with a cut-off point of 60 for high level of perceived stress. The higher the score, the greater the sense of stress. PSQ will be performed at the beginning and after four weeks of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Joanna Szczepańska-Gieracha, Prof., Study Chair — University School of Physical Education in Wroclaw, Poland
Locations (1):
- Foundation for Senior Citizen Activation SIWY DYM, Wroclaw, Lower Silesian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alberti KG, Zimmet P, Shaw J. Metabolic syndrome--a new world-wide definition. A Consensus Statement from the International Diabetes Federation. Diabet Med. 2006 May;23(5):469-80. doi: 10.1111/j.1464-5491.2006.01858.x. PMID 16681555
- [Background] Archer T, Josefsson T, Lindwall M. Effects of physical exercise on depressive symptoms and biomarkers in depression. CNS Neurol Disord Drug Targets. 2014;13(10):1640-53. doi: 10.2174/1871527313666141130203245. PMID 25470398
- [Background] Baert V, Gorus E, Mets T, Geerts C, Bautmans I. Motivators and barriers for physical activity in the oldest old: a systematic review. Ageing Res Rev. 2011 Sep;10(4):464-74. doi: 10.1016/j.arr.2011.04.001. Epub 2011 May 5. PMID 21570493
- [Background] Greenberg SA. How to try this: the Geriatric Depression Scale: Short Form. Am J Nurs. 2007 Oct;107(10):60-9; quiz 69-70. doi: 10.1097/01.NAJ.0000292204.52313.f3. PMID 17895733
- [Background] Hearing CM, Chang WC, Szuhany KL, Deckersbach T, Nierenberg AA, Sylvia LG. Physical Exercise for Treatment of Mood Disorders: A Critical Review. Curr Behav Neurosci Rep. 2016 Dec;3(4):350-359. doi: 10.1007/s40473-016-0089-y. Epub 2016 Oct 14. PMID 28503402
- [Background] Holzel LP, Harter M, Hull M. [Multiprofessional outpatient psychosocial treatment for elderly patients with mental disorders]. Nervenarzt. 2017 Nov;88(11):1227-1233. doi: 10.1007/s00115-017-0407-y. German. PMID 28871311
- [Background] Hsieh PL. A school-based health promotion program for stressed nursing students in Taiwan. J Nurs Res. 2011 Sep;19(3):230-7. doi: 10.1097/JNR.0b013e318228d010. PMID 21857330